CLINICAL TRIAL: NCT03837353
Title: A Parallel Arm Phase 1b/2a Study of DKN-01 as Monotherapy or in Combination With Docetaxel for the Treatment of Advanced Prostate Cancer With Elevated DKK1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated early due to slow accrual in the context of changing practice patterns.
Sponsor: NYU Langone Health (Other)
Collaborators: Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01747
Record Dates: First submitted 2019-01-22; First posted 2019-02-12 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1A (Experimental): In dose-escalation Cohort 1A, the dose of docetaxel 75 mg/m2 will remain fixed. The DKN-01 dose level will start with 300 mg and be escalated to 600 mg or de-escalated to 150 mg depending on the absence or presence of identified DLTs. DKN-01 will be administered in combination with docetaxel on Day 1 and as monotherapy on Day 15 of each 21-day cycle. Patients will be treated with the combination of DKN-01 and Docetaxel until Prostate Cancer Working Group 3 (PCWG3) progression or unacceptable toxicity.
  Interventions: Drug: DKN-01; Drug: Docetaxel
- Cohort 1B (Experimental): In dose-expansion Cohort 1B, either the maximum tolerated dose (MTD) or highest dose tested of DKN-01 in combination with docetaxel in Cohort 1A will be the dose used. The dose of docetaxel 75 mg/m2 will remain fixed. DKN-01 will be administered in combination with docetaxel on Day 1 and as monotherapy on Day 15 of each 21-day cycle. Patients will be treated with the combination of DKN-01 and Docetaxel until PCWG3 progression or unacceptable toxicity.
  Interventions: Drug: DKN-01; Drug: Docetaxel
- Cohort 2A (Experimental): In dose-escalation Cohort 2A, DKN-01 dose level will start with 300 mg and be escalated to 600 mg or de-escalated to 150 mg depending on the absence or presence of identified DLTs. DKN-01 will be administered as monotherapy on Days 1 and 15 of each 28-day cycle. Patients will be treated with DKN-01 until PCWG3 progression or unacceptable toxicity.
  Interventions: Drug: DKN-01
- Cohort 2B (Experimental): In dose-expansion Cohort 2B, the MTD or highest dose tested of DKN-01 monotherapy in Cohort 2A will be the dose used. DKN-01 will be administered as monotherapy on Days 1 and 15 of each 28-day cycle. Patients will be treated with DKN-01 until PCWG3 progression or unacceptable toxicity.
  Interventions: Drug: DKN-01

INTERVENTIONS:
Drug: DKN-01 — DKN-01 is a large molecular weight protein that will be given as a flat dose on a Days 1 and 15 of a 21-day cycle in Dose-Escalation Cohort 1A and Dose-Expansion Cohort 1B. DKN-01 will be given on Days 1 and 15 on a 28-day cycle in Dose-Escalation Cohort 2A and Dose-Expansion Cohort 2B. The dose of DKN-01 will be administered as an intravenous (IV) infusion over 60 (±) 15 minutes.
Drug: Docetaxel — Docetaxel will be administered as an IV infusion over approximately 60 (±15) minutes on day 1 of a 21-day cycle in Cohorts 1A and 1B. In Cohort 1A, docetaxel must be dosed at 75 mg/m2 on cycle 1 day 1. Docetaxel can be dosed at 75 mg/m2 or 60 mg/m2 in subsequent cycles depending on clinical discretion and dose modification guidelines. Regardless of dose, docetaxel must be dosed in 21-day cycles. In Cohort 1B, cycle 1 day 1 dosing of docetaxel will either be 75 mg/m2 or 60 mg/m2 depending on clinical discretion.
  Arms: Cohort 1A; Cohort 1B

SUMMARY:
This is a non-randomized multi-center Phase 1b/2a dose escalation and dose expansion study testing DKN-01 as monotherapy or in combination with docetaxel in metastatic castration-resistant prostate cancer. Patients need to be biomarker positive (Dickkopf-1 [DKK1]) either in plasma or biopsy. Other biopsies for correlative studies are encouraged but not mandatory. Pharmacokinetic (PK) testing of one pre-treatment blood sample and one post-treatment blood sample will be mandatory on Day 1 of every cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Have a histologically or cytologically confirmed cancer of prostate origin (adenocarcinoma, poorly differentiated carcinoma, or neuroendocrine carcinoma are all allowed).

  * Patients with pure neuroendocrine carcinoma must have had at least one line of platinum-based chemotherapy unless the patient is intolerant of or is refusing chemotherapy.
  * Patients with pure neuroendocrine carcinoma do not need to have been previously treated with androgen receptor (AR) signaling inhibitors (abiraterone or enzalutamide or apalutamide or darolutamide) but must have castrate testosterone and have castration-resistant disease.
* Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nM). If the patient is being treated with luteinizing hormone-releasing hormone (LHRH) agonists (patient who have not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to C1D1 and must be continued throughout the study.
* Cohorts 1A, 1B: Patients must have progressed despite 1 or more androgen receptor (AR) signaling inhibitors (abiraterone or enzalutamide or apalutamide or darolutamide) and have not received prior taxane-based chemotherapy for prostate cancer. Prior treatment with an AR signaling inhibitor for castration-sensitive disease will be allowed if the time to progression was within 1 year after starting drug. Prior treatment with a taxane-based chemotherapy for castration-sensitive disease will be exclusionary. (Prior treatment with an AR signaling inhibitor is not required for pure prostate neuroendocrine carcinoma as in inclusion 2.)
* Cohorts 2A and 2B: Patients must have progressed despite 1 or more AR signaling inhibitor (abiraterone or enzalutamide or apalutamide or darolutamide) and either had disease progression, were intolerant of, or refused 1 or more taxane-based chemotherapies for mCRPC. (Prior treatment with an AR signaling inhibitor is not required for pure prostate neuroendocrine carcinoma as in inclusion 2.)
* Cohort 1B. Patients must have measurable disease per RECIST v1.1 guidelines AND must have either:

  * PSA progression is defined by Prostate Cancer Working Group 3 (PCWG3) criteria as a minimum of two consecutive rising levels, with an interval of ≥1 week between each determination with a minimum PSA of 1 ng/mL, if PSA is the sole evidence of progression, OR
  * Radionuclide bone progression as defined by at least two new metastatic lesions (per PCWG3), OR
  * Soft tissue progression on transaxial imaging: new or progressive soft tissue masses on computed tomography (CT) or magnetic resonance imaging (MRI) scans as defined by RECIST v1.1.
* Cohorts 1A, 2A, 2B. Patients must have baseline progression defined as one of the following:

  * PSA progression is defined by PCWG3 criteria as a minimum of two consecutive rising levels, with an interval of ≥1 week between each determination with a minimum PSA of 2 ng/mL.
  * Radionuclide bone progression as defined by at least two new metastatic lesions (per PCWG3).
  * Soft tissue progression on transaxial imaging: new or progressive soft tissue masses on computed tomography (CT) or magnetic resonance imaging (MRI) scans as defined by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Estimated life expectancy of at least 3 months, in the judgment of the Investigator.
* Required initial laboratory values within 14 days of C1D1:

  * Total bilirubin within normal limits for the institution. (For Cohorts 2A and 2B, total bilirubin < 3 × ULN is acceptable with known liver metastases).
  * For Cohorts 1A, 1B transaminases [aspartate aminotransferase (AST) and alanine aminotransferase (ALT)] ≤1.5 × the upper limit of normal (ULN). For Cohorts 2A and 2B, AST and ALT ≤ 5.0 × ULN is acceptable with known liver metastases.
  * Creatinine ≤2.0 or calculated creatinine clearance ≥50 mL/min using the Cockcroft and Gault Method (Cockroft and Gault 1976).
  * Absolute neutrophil count ≥1000 cells/µl.
  * Absolute lymphocyte count ≥500/µl.
  * Hemoglobin ≥8.5 g/dL.
  * Platelet count ≥100,000 cells/µl. (For Cohorts 2A and 2B, Platelet count ≥75,000 cells/µl).
  * International normalized ratio (INR) (prothrombin time [PT])/partial thromboplastin time (PTT) ≤1.5 × ULN unless receiving anticoagulant, in which case INR ≤3.0 and no active bleeding, (ie, no clinically significant bleeding within 14 days prior to first dose of study therapy.
* Sexually active male patients must agree to use adequate contraception (hormonal or barrier method of birth control) during the study and for 6 months after their last dose of study drug. Should a patient's partner become pregnant or suspect she is pregnant while participating in the study, the Investigator should be immediately informed.
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study-specific procedures.
* Provided written informed consent prior to any study-specific procedures.
* Submission of a next-generation sequencing report from prostate cancer tissue or ctDNA from a CLIA certified lab if available. If no such report is available, a statement attesting to the lack of such a report is sufficient for eligibility.

Exclusion Criteria:

* Any anti-cancer therapy (with the exception of luteinizing hormone-releasing hormone [LHRH] analog or antagonist) within 2 weeks prior to initiation of study treatment.
* Any investigational anti-cancer therapy within 4 weeks of initiation of study treatment.
* New York Heart Association Class III or IV heart failure, or myocardial infarction within the past 6 months, or unstable arrhythmia within 3 months.
* Uncontrolled bacterial, viral, or fungal infections, within 7 days of study entry.
* History of malignancy other than prostate cancer within 2 years prior to screening, except for malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as non-melanoma skin carcinoma or ductal carcinoma in situ.
* Known to be human immunodeficiency virus (HIV) positive, have positive hepatitis B surface antigen (HBSAg), or positive hepatitis C antibody (HCAb) test. (Hepatitis C antibody-positive patients with an undetectable hepatitis C virus (HCV) RNA will be eligible.)
* History of solid organ transplant (ie, heart, lungs, liver, or kidney).
* History of autologous/allogenic bone marrow transplant.
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the Investigator and/or Sponsor.
* Major surgical procedures or significant traumatic injury within 4 weeks prior to study entry (minor surgical procedures within 1 week of study entry). Note: Diagnostic cystoscopy is not exclusionary at any time during screening. History of osteonecrosis of the hip. Other hip pathology such as degenerative disease or malignant involvement are not exclusionary. Screening of asymptomatic patients is not required.
* Active or untreated central nervous system (CNS) malignancy or metastasis. Screening for CNS metastases of asymptomatic patients without a history of CNS metastases is not required. Patients with treated CNS metastases are eligible provided they meet all of the following criteria:

  * Evaluable disease outside the CNS.
  * No history of intracranial or intraspinal hemorrhage.
  * No evidence of significant vasogenic edema.
  * No ongoing requirement for corticosteroids as therapy for CNS disease. (Anti-convulsants at a stable dose for > one month is allowed.)
  * No stereotactic radiation, whole brain radiation within 4 weeks of C1D1.
  * Patients with CNS metastases treated by neurosurgical resection or brain biopsy within 3 month prior to C1D1 will not be allowed.
  * Radiographic demonstration of interim stability (ie, no progression) between completion of CNS-directed therapy and the screening radiographic study.
  * Screening CNS radiographic study ≥4 weeks since completion of radiotherapy or surgical resection and ≥2 weeks since discontinuation of corticosteroids.
* Any other condition, disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
* Active substance abuse.
* Receipt of any live vaccine within 30 days before the first dose of study treatment or anticipation that such a live vaccine will be required during study participation.
* Previously treated with an anti-DKK1 therapy.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wise, MD, PhD, Principal Investigator — New York Langone Medical Center
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Veterans Affairs New York Harbor Healthcare System, New York, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.

REFERENCES:
- [Derived] Wise DR, Schneider JA, Armenia J, Febles VA, McLaughlin B, Brennan R, Thoren KL, Abida W, Sfanos KS, De Marzo AM, Yegnasubramanian S, Fox JJ, Haas M, Heath H, Kagey MH, Newman W, Sirard CA, Fleisher M, Morris MJ, Chen Y, Larson SM, Haffner MC, Nelson PS, Schultz N, Garabedian MJ, Scher HI, Logan SK, Sawyers CL; International SU2C/PCF Prostate Cancer Dream Team. Dickkopf-1 Can Lead to Immune Evasion in Metastatic Castration-Resistant Prostate Cancer. JCO Precis Oncol. 2020 Sep 29;4:PO.20.00097. doi: 10.1200/PO.20.00097. eCollection 2020. PMID 33015525

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1A.1 (DKN-01 300mg, Docetaxel 75 mg/m2): Participants in the dose-escalation Cohort 1A.1 who received DKN-01 300mg and Docetaxel 75 mg/m2.
- Cohort 1A.2 (DKN-01 600mg, Docetaxel 75 mg/m2): Participants in the dose-escalation Cohort 1A.2 who received DKN-01 600mg and Docetaxel 75 mg/m2.
- Cohort 1B (DKN-01 600mg [Phase II Dose], Docetaxel 75 mg/m2): Participants in the Phase II dose-expansion Cohort 1B who received DKN-01 600mg [Phase II Dose] and Docetaxel 75 mg/m2.
- Cohort 2A.1 (DKN-01 300mg): Participants in dose-escalation Cohort 2A.1 who received DKN-01 300mg monotherapy.
- Cohort 2A.2 (DKN-01 600mg): Participants in dose-escalation Cohort 2A.1 who received DKN-01 600mg monotherapy.
- Cohort 2B (DKN-01 600mg [Phase 2 Dose]): Participants in the Phase II dose-expansion Cohort 2B who received DKN-01 600mg [Phase II Dose] monotherapy.
Period: Overall Study
Arm/Group | Cohort 1A.1 (DKN-01 300mg, Docetaxel 75 mg/m2) | Cohort 1A.2 (DKN-01 600mg, Docetaxel 75 mg/m2) | Cohort 1B (DKN-01 600mg [Phase II Dose], Docetaxel 75 mg/m2) | Cohort 2A.1 (DKN-01 300mg) | Cohort 2A.2 (DKN-01 600mg) | Cohort 2B (DKN-01 600mg [Phase 2 Dose])
Started | 3 | 3 | 2 | 4 | 3 | 3
Completed | 3 | 3 | 2 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1A.1 (DKN-01 300mg, Docetaxel 75 mg/m2) | Cohort 1A.2 (DKN-01 600mg, Docetaxel 75 mg/m2) | Cohort 1B (DKN-01 600mg [Phase II Dose], Docetaxel 75 mg/m2) | Cohort 2A.1 (DKN-01 300mg) | Cohort 2A.2 (DKN-01 600mg) | Cohort 2B (DKN-01 600mg [Phase 2 Dose]) | Total
Number analyzed (Participants) | 3 | 3 | 2 | 4 | 3 | 3 | 18
Age, Continuous [Median (Full Range); unit: years] | 66 [59 to 67] | 68 [67 to 71] | 76 [72 to 80] | 65 [57 to 83] | 74 [72 to 78] | 64 [60 to 65] | 70 [57 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 2 | 4 | 3 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 3 | 0 | 4 | 3 | 2 | 14
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 1 | 0 | 3
  White | 2 | 3 | 2 | 2 | 2 | 2 | 13
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 | 4 | 3 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities Observed by End of Treatment Cycle 1
Description: Measured among Phase I dose-escalation cohorts (arms 1A.1, 1A.2, 2A.1, and 2A.2) only.
Time Frame: Up to End of Cycle 1 (Up to Day 21 for Cohort 1A, Up to Day 28 for Cohort 2A)
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Cohort 1A.1 (DKN-01 300mg, Docetaxel 75 mg/m2) | Cohort 1A.2 (DKN-01 600mg, Docetaxel 75 mg/m2) | Cohort 2A.1 (DKN-01 300mg) | Cohort 2A.2 (DKN-01 600mg)
Number analyzed (Participants) | 3 | 3 | 4 | 3
Number of events | 0 (0) | 0 (0) | 0 (0) | 0 (0)

2. Primary Outcome: Number of Participants With a Best Overall Response of Complete Response (iCR) or Partial Response (iPR) Per iRECIST by End of Long-Term Follow-Up Period
Description: iRECIST will be used by the Investigator to assess tumor response and progression. An iCR is defined as the disappearance of all target lesions as assessed by iRECIST; an iPR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters, as assessed by iRECIST.
Time Frame: Up to Year 2 Post-Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A.1 (DKN-01 300mg, Docetaxel 75 mg/m2) | Cohort 1A.2 (DKN-01 600mg, Docetaxel 75 mg/m2) | Cohort 1B (DKN-01 600mg [Phase II Dose], Docetaxel 75 mg/m2) | Cohort 2A.1 (DKN-01 300mg) | Cohort 2A.2 (DKN-01 600mg) | Cohort 2B (DKN-01 600mg [Phase 2 Dose])
Number analyzed (Participants) | 3 | 3 | 2 | 4 | 3 | 3
Participants | 3 | 2 | 0 | 0 | 0 | 0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Defined as the time from the first dose of study treatment to documentation of radiographic progression in soft tissue as assessed by Investigator using iRECIST, in bone as assessed by Investigator using Prostate Cancer Working Group 3 (PCWG3), or death, whichever occurs first.
Time Frame: Up to Year 2 Post-Baseline
Population: Data for this outcome measure was not collected among participants in the Monotherapy arms (2A.1, 2A.2, and 2B).
Measure: Median (Full Range); unit: Months
Arm/Group | Cohort 1A.1 (DKN-01 300mg, Docetaxel 75 mg/m2) | Cohort 1A.2 (DKN-01 600mg, Docetaxel 75 mg/m2) | Cohort 1B (DKN-01 600mg [Phase II Dose], Docetaxel 75 mg/m2) | Cohort 2A.1 (DKN-01 300mg) | Cohort 2A.2 (DKN-01 600mg) | Cohort 2B (DKN-01 600mg [Phase 2 Dose])
Number analyzed (Participants) | 3 | 3 | 2 | 0 | 0 | 0
Months | 6.3 [5.1 to 6.6] | 8.1 [4.2 to 8.5] | 2 [1.2 to 2.7] |  |  |

4. Secondary Outcome: Number of Participants With a Decline in Prostate-Specific Antigen (PSA) of at Least 50% Relative to Baseline
Time Frame: Up to Year 2 Post-Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1A.1 (DKN-01 300mg, Docetaxel 75 mg/m2) | Cohort 1A.2 (DKN-01 600mg, Docetaxel 75 mg/m2) | Cohort 1B (DKN-01 600mg [Phase II Dose], Docetaxel 75 mg/m2) | Cohort 2A.1 (DKN-01 300mg) | Cohort 2A.2 (DKN-01 600mg) | Cohort 2B (DKN-01 600mg [Phase 2 Dose])
Number analyzed (Participants) | 3 | 3 | 2 | 4 | 3 | 3
Participants | 3 | 2 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximal Percent Change in PSA Measured After Treatment Initiation
Time Frame: Up to Year 2 Post-Baseline
Measure: Median (Full Range); unit: Percentage
Arm/Group | Cohort 1A.1 (DKN-01 300mg, Docetaxel 75 mg/m2) | Cohort 1A.2 (DKN-01 600mg, Docetaxel 75 mg/m2) | Cohort 1B (DKN-01 600mg [Phase II Dose], Docetaxel 75 mg/m2) | Cohort 2A.1 (DKN-01 300mg) | Cohort 2A.2 (DKN-01 600mg) | Cohort 2B (DKN-01 600mg [Phase 2 Dose])
Number analyzed (Participants) | 3 | 3 | 2 | 4 | 3 | 3
Percentage | -74 [-94 to -57] | -87 [-100 to -23] | 0 [-45 to 40] | 93 [-8 to 317] | 57 [6 to 78] | 28 [17 to 174]

ADVERSE EVENTS:
Time Frame: 40 months
Description: PI to monitor for AEs at every follow-up visit.
Groups:
- DKN-01 300mg, Docetaxel 75 mg/m2: Participants who received DKN-01 300mg and Docetaxel 75 mg/m2.
- DKN-01 600mg, Docetaxel 75 mg/m2: Participants who received DKN-01 600mg and Docetaxel 75 mg/m2.
- DKN-01 300mg: Participants who received DKN-01 300mg monotherapy.
- DKN-01 600mg: Participants who received DKN-01 600mg monotherapy.
Arm/Group | DKN-01 300mg, Docetaxel 75 mg/m2 | DKN-01 600mg, Docetaxel 75 mg/m2 | DKN-01 300mg | DKN-01 600mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/5 | 0/4 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DKN-01 300mg, Docetaxel 75 mg/m2 (N=3) | DKN-01 600mg, Docetaxel 75 mg/m2 (N=5) | DKN-01 300mg (N=4) | DKN-01 600mg (N=6)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Clostridium Difficile (Serious Adverse Event) (Infections and infestations) | 1 | 0 | 0 | 0
Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DKN-01 300mg, Docetaxel 75 mg/m2 (N=3) | DKN-01 600mg, Docetaxel 75 mg/m2 (N=5) | DKN-01 300mg (N=4) | DKN-01 600mg (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1
alanine transaminase (ALT) levels increased (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Alkaline Phosphatase (ALP) Levels Increased (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Alopecia (General disorders) | 3 | 2 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Anorexia (General disorders) | 0 | 2 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Aspartate aminotransferase (AST) levels increased (Hepatobiliary disorders) | 0 | 2 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 4
Blood bilirubin increased (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Blurred Vision (Eye disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cardiac disorders (Cardiac disorders) | 0 | 1 | 1 | 0
Chills (General disorders) | 0 | 2 | 0 | 0
Confusion (Nervous system disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 2
Creatine phosphokinase (CPK) levels increased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Creatinine increased (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dehydration (General disorders) | 2 | 1 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Dysgeusia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Edema limbs (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Epistaxis (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Fall (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 4 | 3 | 3
Fecal Incontinence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Gait disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Gastroeosphgeal Reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal Disorders (Gastrointestinal disorders) | 1 | 1 | 0 | 0
General Disorders and Administrative Site Condition (General disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 2
Hypertension (Cardiac disorders) | 0 | 1 | 0 | 0
Hypoalbuminemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hypocalcemia (Renal and urinary disorders) | 0 | 1 | 0 | 1
Hypokalemia (Renal and urinary disorders) | 1 | 1 | 0 | 0
Hypomagnesemia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hypotension (Cardiac disorders) | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 1
Infusion related reaction (General disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1
Insomnia (General disorders) | 0 | 2 | 0 | 1
Localized edema (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Mucositis oral (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal/connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 1 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Nervous system disorders (Nervous system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Penile infection (Infections and infestations) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 0 | 2
Phlebitis (Vascular disorders) | 1 | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pruritus (General disorders) | 0 | 2 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
Rectal mucositis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Renal and urinary disorders (Renal and urinary disorders) | 1 | 0 | 1 | 0
Surgical and Medical procedure (General disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 1 | 0
Vascular Disorder (Vascular disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Watering eyes (Eye disorders) | 0 | 1 | 0 | 0
White Blood Cells Decreased (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT03837353/Prot_SAP_000.pdf